CLINICAL TRIAL: NCT03455842
Title: International Multicenter Comparative Randomized Double-blind Placebo-controlled Clinical Study of Efficacy and Safety of BCD-089 in Different Dosing Regimens in Patients With Active Rheumatoid Arthritis
Brief Title: The BCD-089 (aIL6R) in Patients With Active Rheumatoid Arthritis
Acronym: AURORA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCD-089-2
Record Dates: First submitted 2018-02-22; First posted 2018-03-07 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2019-12

CONDITIONS: Seropositive RA
MeSH Terms: interventions — levilimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BCD-089 weekly (Experimental)
  Interventions: Biological: BCD-089, 162 mg, s/c, qw
- BCD-089 biweekly (Experimental)
  Interventions: Biological: BCD-089, 162 mg, s/c, q2w
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Biological: BCD-089, 162 mg, s/c, qw — Subcutaneous injections of anti-IL6R every week
  Arms: BCD-089 weekly
Biological: BCD-089, 162 mg, s/c, q2w — Subcutaneous injections of anti-IL6R every other week
  Arms: BCD-089 biweekly
Drug: placebo — Subcutaneous injections of placebo every week, until week 12. Thereafter subcutaneous injections of anti-IL6R every other week
  Arms: Placebo

SUMMARY:
The study is Phase II randomized, double-blind, placebo-controlled clinical trial to evaluate efficacy and safety, pharmacokinetics and pharmacodynamics of 2 dosing regimens (qw and q2w, s/c) of monoclonal antibody to IL6R (BCD-089) in patients with active rheumatoid arthritis and inadequate response to methotrexate.

DETAILED DESCRIPTION:
IL-6 is a new potential therapeutic target which plays important role in pathogenesis of several autoimmune disorders including rheumatoid arthritis. BCD-089 is a novel fully human monoclonal antibody against the interleukin-6 receptor developed by JCS BIOCAD (Russia) which is successfully passed phase I clinical study. Fixed dose of 162 mg was chosen for evaluation in phase II clinical trial. Comparisons in terms of efficacy, safety, PK/PD will be made for every week and every other week dosing for 54 weeks. W0-W12, planed as blinded, "main" period of the study, consists of three arms (n=35, each) - 2 study arms and placebo arm and served to test the hypothesis of superiority of BCD-089 to placebo. W12-W54, planned as "open" period of the study and served to evaluate long-therm safety and efficacy of BCD-089 in patients with active rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Males and females aged 18 - 80 years, at IC signing date.
3. Diagnosis of rheumatoid arthritis, according to ACR 2010 criteria, at least for 6 month prior to IC signing date.
4. Active rheumatoid arthritis at IC signing date.
5. Therapy with methotrexate for at least 3 month prior to IC signing date.
6. Stable dose of methotrexate (10-25 mg/week) for 4 weeks prior to IC signing date.
7. Persistent activity of RA despite methotrexate (provided by Sponsor) therapy within screening period (4-6weeks).
8. Patients, with following parameters of laboratory investigations:

   • Hemoglobin ≥ 80 g/l;
   * White blood cells ≥ 3,0×109/l;
   * Platelets ≥ 100×109/l;
   * Neutrophils ≥ 2×109/l;
   * ALT and AST < 1,5 × UNL (according to the local / central laboratory normal values)
   * Serum creatinine < 1,7 × UNL (according to the local / central laboratory normal values)
9. Negative urine pregnancy test for women at screening (only for women with childbearing potential - not applied to women at menopause for at least 2 years or surgically sterilized).
10. Patients ability to follow the protocol procedures (according to PI opinion)
11. Patient and his/her sexual partner with childbearing potential are ready to use reliable contraception, starting at the date of IC sign, within the study period and 4 weeks after the last dose of investigational drug administration. (Not applied to participants/sexual partners who surgically sterilized, and women at menopause for more than 2 years). Reliable contraception considered as 1 barrier method and one of the following: spermicides, oral contraception or intrauterine devices)

Exclusion Criteria:

* 1. History of therapy with tocilizumab or other monoclonal antibodies to IL6R / IL6.

  2. History of therapy with rituximab or other B-cell depleting medicines. 3. Felty's syndrome (any form). 4. ACR1991 functional status IV. 5. Low disease activity of rheumatoid arthritis (DAS28-CRP(4) < 3,2). 6. Known allergy or intolerance of any investigational drug/placebo ingredients.

  7. Concomitant medication including any of the following:

  • Requirement > 10 mg / day of oral prednisolone (or equivalent);
  * Requirement < 10 mg / day of oral prednisolone (or equivalent), if the dose was not stable for 4 weeks prior the date of informed consent sign (it is allowed to include patients on topical steroids);
  * Requirement of NSAID, if dose was not stable for 4 weeks prior the date of informed consent sign (it is allowed to include patients received NSAID occasionally to treat intercurrent fever or allergy).
  * Intake of alkalizing agents at any time during 12 month prior the date of IC sign.
  * Intraarticular administration of steroids within 4 month prior the date of IC sign
  * Vaccination with live or attenuated vaccines at any time during 8 weeks preceding the date of IC sign 8. Leflunomide intake within 8 weeks prior the date of IC sign. 9. Therapy with TNF inhibitors, JAK-inhibitors, T-lymphocyte co-stimulation blockers within 2 month prior to the date of IC sign.

    10. Diagnosis or history of severe immunodeficiency. 11. HIV, HCV, HBV, Syphilis. 12. Diagnosis or history of tuberculosis. 13. Latent TB (positive Diaskin test® or QuantiFERON®-TB Gold or T-SPOT.TB or Mantoux/PPD with lack of TB signs on chest X-ray).

    14. It is allowed to include patients with inconclusive Diaskin test® or QuantiFERON®-TB Gold or T-SPOT.TB or Mantoux/PPD, providing that TB has been ruled out (and documented) by TB-specialist (Phtisyatrician) 15. It is allowed to include patients with positive Mantoux/PPD with no signs of TB on chest X-ray, providing that Diaskin test® or QuantiFERON®-TB Gold or T-SPOT.TB was additionally made with negative results and TB has been ruled out (and documented) by TB-specialist (Phtisyatrician) 16. History of Herpes Zoster. 17. Documented chicken pox within 30 days prior to IC sign 18. Diagnosis of any other chronic infection (sepsis, invasive mycosis, histoplasmosis etc.), which may increase the risk of infectious adverse events.

    19. Any acute infection or chronic infection flare within 30 days prior to informed consent sign, which may increase (according to the PI opinion) the risk of infectious adverse events.

    20. Severe infections (required hospitalization, systemic antimicrobial/antifungal/antiviral treatment) within 6 months prior to date of IC sign.

    21. Systemic antimicrobial, antifungal, antiviral or anthelminthic medication within 2 months prior to fate of IC date.

    22. More than 4 cases of acute respiratory infections within 6 month prior to IC date.

    23. Major surgical interventions within 30 days prior to IC date or planned surgical intervention within the period of the study participation.

    24. History of seizures. 25. History of depression, suicidal ideation/behavior. 26. Diverticulosis or diverticulitis. 27. Known history of alcohol or drug abuse, or signs of alcohol/drug dependence at present time, which according to the PI opinion could interfere with RA treatment or reduce compliance.

    28. Any other documented conditions which increase the risk of AEs development or may interfere with symptoms of RA (masking, increasing or changing) or induce clinical symptoms or laboratory abnormalities similar to RA:
    1. Uncontrolled diabetes mellitus;
    2. Severe, uncontrolled hypertonia;
    3. Presence or history of inflammatory joint disease other than RA (ankylosing spondylitis, gout, psoriatic arthritis, Lyme disease) or any other systemic autoimmune disease (including lupus, Crohn's disease, ulcerative colitis, scleroderma, inflammatory myopathy, mixed connective tissue disease, autoimmune overlap syndrome, fibromyalgia etc.);
    4. Any history of malignancy, excluding cured basal cell carcinoma / cervical cancer in situ (complete remission for 5 years); cured basal cell skin carcinoma (5 years complete remission), cured ductal breast cancer (5 years complete remission);
    5. Decompensated liver or kidney diseases;
    6. Unstable angina pectoris;
    7. Chronic heart failure, class III-IV according to NYHA;
    8. Myocardial infarction, within 1 year prior to IC sign;
    9. History of organ transplantation;
    10. History of Quincke edema; History of any significant respiratory diseases, including COPD, asthma or bronchiectasis disease;
    11. Decompensated respiratory failure;
    12. History of multiple sclerosis, Devic's disease, or Guillain-Barre syndrome;
    13. Any neurological disease with motor or sensory functions impairment. 29. Pregnancy, current or planned in less than 8 weeks after study completion or breastfeeding.

        30. Simultaneous participation in other clinical trials or participation in other clinical trials with 3 month prior to IC signing date or history of participation it current clinical study (excluding patients dropped out at screening).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-10-22 (Actual)

PRIMARY OUTCOMES:
ACR20 | week 12

SECONDARY OUTCOMES:
ACR50 | week 4, week 8, week 16, week 24, week 36, week 48, week 52
ACR70 | week 4, week 8, week 16, week 24, week 36, week 48, week 52
Low RA activity | week 4, week 8, week 12, week 16, week 24, week 36, week 48, week 52
  DAS28-CRP(4)<3.2
Low RA activity | week 4, week 8, week 12, week 16, week 24, week 36, week 48, week 52
  SDAI = 11 or less
Low RA activity | week 4, week 8, week 12, week 16, week 24, week 36, week 48, week 52
  CDAI = 10 or less
RA remission | week 24, week 36, week 48, week 52
  According to the ACR/EULAR 2011 remission criteria
X-ray signs of RA | week52
Pharmacokinetics of BCD-089 | week 0 - week 12
  Area Under the BCD-089 Plasma Concentration Versus Time Curve [AUC0-last]
Pharmacokinetics of BCD-089 | week 0 - week 12
  Peak Plasma Concentration [Cmax]
Pharmacokinetics of BCD-089 | week 0 - week 12
  Minimum Plasma Concentration [Cmin]
Pharmacokinetics of BCD-089 | week 0 - week 12
  Time to Maximum Plasma Concentration [Tmax]
Pharmacokinetics of BCD-089 | week 0 - week 12
  Time to Minimum Plasma Concentration [Tmin]
Pharmacokinetics of BCD-089 | week 0 - week 12
  Accumulation Ratio [AR]
Pharmacodynamics of BCD-089 | week 0 - week 12
  Plasma concentration of CRP
Pharmacodynamics of BCD-089 | week 0 - week 12
  Plasma concentration of Interleukin-6
Pharmacodynamics of BCD-089 | week 0 - week 12
  Plasma concentration of soluble receptor of interleukin-6
Pharmacodynamics of BCD-089 | week 0 - week 12
  Plasma concentration of tumor necrosis factor - alpha

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ivanov, PhD, Study Chair — Biocad
Locations (4):
- 1st City Clinical Hospital, Minsk, Belarus
- Russia (3):
  - Chelyabinsk Regional Clinical hospital, Chelyabinsk
  - Kazan State Medical University, Kazan'
  - North-Western State Medical University n.a. I.I.Mechnikov, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mazurov V.I., Korolev M.A., Prystrom A.M., Kunder E.V., Soroka N.F., Kastanayan A.A., Povarova T.V., Plaksina T.V., Antipova O.V., Kretchikova D.G., Smakotina S.A., Tciupa O.A., Puntus E.V., Raskina T.A., Shilova L.N., Kropotina T.V., Nesmeyanova O.B., Popova T.A., Vinogradova I.B., Linkova Yu.N., Dokukina E.A., Plotnikova A.V., Pukhtinskaia P.S., Zinkina-Orikhan A.V., Eremeeva A.V., Lutckii A.A. Effectiveness and safety of levilimab in combination with methotrexate in treatment of patients with active rheumatoid arthritis resistant to methotrexate monotherapy (double-blinded randomized placebo controlled phase III clinical study SOLAR). Modern Rheumatology Journal. 2021;15(4):13-23. https://doi.org/10.14412/1996-7012-2021-4-13-23
- See also: Related Info — https://mrj.ima-press.net/mrj/article/view/1164/1169